CLINICAL TRIAL: NCT06383169
Title: Impact of External Drainage of the Lumbar Cistern in Patients With Hydrocephalus Following Meningioma Surgery and Its Influence on Patient Satisfaction
Status: Completed | Type: Observational
Sponsor: First Hospital of Zhangjiakou City (Other)
Responsible Party: Sponsor
Other Study IDs: wanglizhong
Record Dates: First submitted 2024-04-22; First posted 2024-04-25 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Investigate the Effect of External Lumbar Cistern Drainage in Preventing Postoperative Hydrocephalus in Patients Who Have Undergone Meningioma Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- observation group
- control group

SUMMARY:
This study aims to investigate the effect of external lumbar cistern drainage in preventing postoperative hydrocephalus in patients who have undergone meningioma surgery and its impact on patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of meningiomas based on established diagnostic criteria and pathological confirmation
* postoperative development of hydrocephalus, specifically communicating hydrocephalus
* absence of other intracranial tumours or contraindications for surgery

Exclusion Criteria:

* concurrent mental disorders, coagulation dysfunction or organic diseases affecting other areas
* hematologic diseases, severe liver or kidney dysfunction
* patients discontinuing treatment or transferring to a higher-level hospital
* a history of hydrocephalus, such as obstructive hydrocephalus

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This retrospective study analysed data from 86 patients who developed postoperative hydrocephalus following meningioma surgery, conducted between May 2019 and May 2022. Based on the inclusion and exclusion criteria, patients were divided into two groups. The control group (n = 43) received conventional treatment methods, and the observation group (n = 43) underwent external drainage of the lumbar cistern.
Sampling Method: Non-Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-30 (Actual)

PRIMARY OUTCOMES:
Comparison of general clinical data | 2 weeks
Comparison of the response rate | 2 weeks
Comparison of GCS scores and intracranial pressure | 2 weeks
Comparison of KPS scores and satisfaction | 2 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- First Hospital of Zhangjiakou City, Zhangjiakou, China